CLINICAL TRIAL: NCT04881045
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY EVALUATING THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND ANTITUMOR ACTIVITY OF PF-07257876 IN PATIENTS WITH ADVANCED OR METASTATIC TUMORS
Brief Title: Study to Test the Safety and Tolerability of PF-07257876 in Participants With Selected Advanced Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4401001; 2022-003338-38 (EudraCT Number)
Record Dates: First submitted 2021-04-09; First posted 2021-05-11 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Non-Small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck; Ovarian Cancer
Keywords: PD-L1 (Programmed death-ligand 1); CD47 (cluster of differentiation 47); immunotherapy; macrophage checkpoint inhibitor; advanced solid tumor; metastatic solid tumor; Ovarian Cancer; Lung Cancer; Non-small cell lung cancer; Head and Neck cancer; SCCHN; NSCLC; solid tumor; advanced cancer; metastatic cancer; Squamous cell carcinoma of the head and neck; Squamous cell head and neck cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Ovarian Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Part 1) (Experimental): Participants will receive PF-07257876 at escalating dose levels.
  Interventions: Biological: PF-07257876
- Dose Expansion (Part 2) - Cohort 1 (NSCLC) (Experimental): Participants with non-small cell lung cancer (NSCLC) will receive PF-07257876 at the recommended dose from Part 1.
  Interventions: Biological: PF-07257876
- Dose Expansion (Part 2) - Cohort 2 (SCCHN) (Experimental): Participants with squamous cell carcinoma of the head and neck (SCCHN) will receive PF-07257876 at the recommended dose from Part 1.
  Interventions: Biological: PF-07257876

INTERVENTIONS:
Biological: PF-07257876 — CD47-PDL-1 bispecific antibody

SUMMARY:
This is a first-in-human, Phase 1, open label, multicenter, multiple dose, dose escalation and dose expansion study intended to evaluate the safety, pharmacokinetic, pharmacodynamic and potential clinical benefit of PF-07257876, a CD47-PD-L1 bispecific antibody, in participants with selected advanced or metastatic tumors for whom no standard therapy is available. The study contains 2 parts, single agent Dose Escalation (Part 1) to determine the recommended dose of PF-07257876, followed by Dose Expansion (Part 2) in selected tumor types at the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of selected advanced or metastatic tumor
* Prior treatment with PD-1 (Programmed cell death 1) or PD-L1 (programmed death-ligand 1) in NSCLC and SCCHN or platinum-based therapy in Ovarian cancer
* Confirmed radiographic progression of disease
* PD-L1 IHC positivity ≥1%
* Have ≥1 measurable lesion as defined by RECIST 1.1 that has not been previously irradiated
* Eastern Cooperative Oncology Group performance status 0-1
* Adequate hematologic, renal and liver functions
* Resolved acute effects of any prior therapy
* Participants in Part 1 must be able to provide archival tumor tissue collected within the prior 6 months or consent to undergo a fresh biopsy during screening. Participants enrolled to the MTD (Maximum Tolerated Dose) cohort in Part 1 must consent to mandatory paired pre-treatment and on-treatment biopsies. Participants in Part 2 must consent to a pre-treatment biopsy and a subset of patients must consent to a paired on-study biopsy as well until the Sponsor deems an adequate number have been received.

Exclusion Criteria:

* Participants with known brain metastasis larger than 4 cm or that is symptomatic. New brain metastases detected at screening. Participants with previously diagnosed brain metastases are eligible if they have completed treatment and recovered from acute effects prior to study entry.
* Abnormal neurological assessment by investigator
* Other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Major surgery or radiation therapy within 4 weeks prior to planned first dose
* Last systemic anti-cancer therapy within 28 days or 5 half-lives (whichever is shorter) prior to planned first dose (6 weeks for mitomycin C or nitrosoureas)
* Active bleeding disorder in the past 6 months prior to first dose
* History of clinically significant severe immune mediated adverse event that was considered related to prior immune modulatory therapy and required immunosuppressive therapy (other than hormone replacement therapy)
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (ie, bronchiolitis obliterans, cryptogenic organizing pneumonia), evidence of active pneumonitis on screening chest CT(computer tomography) scan
* Anticoagulation with vitamin K antagonists or factor Xa inhibitors is not allowed
* Treatment with chronic systemic corticosteroids or other immunosuppressive medications
* Participation in other studies involving investigational drug(s) within 4 weeks prior to planned first dose
* Active, uncontrolled bacterial, fungal, or viral infection, Hepatitis B, Hepatitis C, or Human immunodeficiency virus (HIV) infection
* Active COVID-19/SARS-CoV2
* Pregnant or breastfeeding female participant
* Organ transplant requiring immunosuppressive treatment or prior allogeneic bone marrow or hematopoietic stem cell transplant
* Significant cardiac or pulmonary conditions or events within previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) in Dose Escalation (Part 1) | Baseline through end of Cycle 1 (each cycle is 28 days)
  DLTs will be evaluated during Cycle 1 (a cycle is 28 days) in Part 1. The number of DLTs will be used to determine the optimal dose
Number of participants with adverse events (AEs) | Baseline through up to 2 years
  AEs characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0), timing, seriousness, and relationship to study therapy.
Number of participants with clinically significant laboratory abnormalities | Baseline through up to 2 years
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Objective response rate (ORR) in the Expansion cohorts (Part 2) | Baseline through up to 2 years or until disease progression
  Tumor response based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Single dose Pharmacokinetics (PK) parameter: Maximal concentration (Cmax) in Part 1 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Maximum observed plasma concentration of PF-07257876 (Cmax)
Single dose PK parameter: Time to maximal plasma concentration (Tmax) in Part 1 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Time to maximal observed plasma concentration of PF-07257876 (Tmax)
Single dose PK parameter: Area under the Curve (AUClast) in Part 1 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Area under the concentration-time curve from time zero to the last quantifiable time point prior to the next dose.
Multiple dose PK parameter: Maximal concentration (Cmax, ss) in Part 1 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Maximum observed steady state plasma concentration of PF-07257876 (Cmax, ss)
Multiple dose PK parameter: Time to maximal plasma concentration (Tmax, ss) in Part 1 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Time to reach Maximum Observed Steady State Plasma Concentration (Tmax,ss).
Multiple dose PK parameter: Area under the Curve (AUCtau, ss) in Part 1 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Area Under the curve within one dose interval at steady state (AUCtau,ss)
Immunogenicity of PF-07257876 | Cycle 1, Cycle 2, Cycle 3, Cycle 4, and pre-dose on Day 1 at Cycle 5 and every third cycle thereafter (all cycles are 28 days) and at End of Treatment, up to 2 years
  Incidence, titers, and duration (if data permit) of antidrug antibodies (ADA) and neutralizing antibodies against PF-07257876
Intratumor T cell levels | Baseline through Cycle 2 Day 15 (each cycle is 28 days)
  Immune biomarker levels in archival biopsies and/or de novo and on-treatment tumor biopsies.
Intratumor PD-L1 expression | Baseline through Cycle 2 Day 15 (each cycle is 28 days)
  PD-L1 expression levels in pretreatment tumor biopsies
ORR in Dose Escalation (Part 1) | Baseline through up to 2 years or until disease progression
  Tumor response assessment based on RECIST 1.1
Duration of response (DOR) | Baseline through up to 2 years or until disease progression
  DOR as assessed using RECIST 1.1
Progression free survival (PFS) | Baseline through up to 2 years or until disease progression
  PFS as assessed using RECIST 1.1
Time to progression (TTP) | Baseline through up to 2 years or until disease progression
  TTP as assessed using RECIST 1.1
Lowest concentration (Ctrough) reached before the next dose is administered in Part 2 | Pre-dose on Day 1 at Cycles 1, 2, 3, 4, 5 and every third cycle thereafter (each cycle is 28 days) and End of Treatment visit, up to 2 years
  PK assessment for PF-07257876
Overall Survival (OS) in the Expansion Cohorts (Part 2) | Baseline through up to 2 years or until disease progression
  Proportion of patients alive

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (39):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Hoag Hospital Irvine, Irvine, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - Keck School of Medicine of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Keck Hospital of USC Pasadena, Pasadena, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate (Emergency Back-Up Only), Santa Monica, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center-North County, Florissant, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Duke Cancer Institute, Durham, North Carolina
  - UPMC Hillman Cancer Center - Camp Hill, Camp Hill, Pennsylvania
  - UPMC Hillman Cancer Center - Carlisle, Carlisle, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Pinnacle - Community Osteopathic / Medical Sciences Pavilion (MSP), Harrisburg, Pennsylvania
  - UPMC Pinnacle - Ortenzio Cancer Center (OCC), Mechanicsburg, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Clinico de Valencia, Valencia, Valenciana, Comunitat

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4401001